CLINICAL TRIAL: NCT03045081
Title: PainTracker Self-Manager: Development and Testing of a Web-based Platform to Promote and Track Chronic Pain Self-management and Other Treatment Outcomes
Brief Title: PainTracker Self-Manager: a Web-based Platform to Promote and Track Chronic Pain Self-management
Acronym: PTSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Duke University (Other); University of New Mexico (Other)
Responsible Party: Principal Investigator, Mark Sullivan, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 51541
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients receive outcome tracking tool, PainTracker, but no additional web-based support for self-management
- PainTracker Self-Manager (Experimental): Patients are invited to complete the web-based PainTracker Self-Manager and interact with a nurse care manager who supports chronic pain self-management
  Interventions: Behavioral: PainTracker Self-Manager

INTERVENTIONS:
Behavioral: PainTracker Self-Manager — Interactive web-based educational and assessment program supported by a nurse care manager
  Arms: PainTracker Self-Manager

SUMMARY:
To develop and test a web-based patient empowerment platform, PainTracker Self-Manager (PTSM), that can support integrated multimodal care in a variety of specialty and primary care settings. The investigators will adapt PainTracker, a web-based outcome and treatment tracking tool already deployed in multiple University of Washington clinics to create the PTSM self-management tool that helps assess, engage, activate, and support patients' efforts to self-manage their chronic pain in collaboration with their clinicians. PTSM design will be based on 4-phase patient engagement strategy derived from Acceptance and Commitment Therapy. Phase 1 focuses on achieving consensus on the clinical problem definition, treatment goals and timeline. Phase 2 focuses on promoting values-based action and acceptance of pain. Phase 3 focuses on providing skills in chronic pain self-management with close monitoring of patient reported outcomes and actigraphy. Phase 4 focuses on providing autonomy support to promote maintenance of self-management behaviors. Phase 5 involves generating a patient registry with the above data for use in quality improvement research. The investigators will engage patients, providers and investigators in designing PTSM, reviewing prototypes, and conducting usability testing. In a 6-month clinical trial, the investigators will compare 50 intervention patients from the UW Center for Pain Relief who receive PTSM to 50 historical control patients who have received the basic PainTracker. The primary outcome will be chronic pain self-efficacy, with secondary outcomes of: chronic pain acceptance, perceived efficacy in physician-patient interactions, and patient and provider satisfaction. Development of the PTSM platform will support the dissemination of the multimodal interdisciplinary care for chronic pain that is recommended in the National Pain Strategy, and may help chronic pain care meet the goals of the Triple Aim: better patient experience, better patient outcomes, with lower costs.

DETAILED DESCRIPTION:
Patients and Setting Study participants (N = 99) were patients seeking care for various chronic pain conditions at the UW CPR between April 2016 and March 2017. The target population for the study was patients who had received an initial treatment planning visit, but who were still early in their course of treatment. Therefore, to be eligible for this study, patients were required to have visited the UW CPR at least once, but not more than 5 times. The control subjects were recruited between April 2016 and September 2016 while the intervention was being developed.The intervention subjects were recruited between September 2016 and March 2017. This sequential, nonrandomized design was chosen because of the limited budget and time available for the development and testing of our intervention.

Measures Demographic and clinical data were extracted from UW CPR electronic medical records. Demographic data collected at enrollment included age, sex, race, ethnicity, and insurance type. Clinical data collected on control and intervention subjects included pain diagnoses, previous and current interventional treatments and therapies for pain,as well as current pain and related medications (opioids, anticonvulsants, antidepressants, anxiolytics, antihistamines, and nonsteroidal anti-inflammatory drugs.

The Pain Self-Efficacy Questionnaire24,25 is a 10-item survey that assesses patients' pain self-efficacy, or confidence in their ability to cope with their pain and continue activities of daily living (eg, "I can cope with my pain in most situations."). Items are scored on a 7-point scale from 0 "not at all confident" to 10 "completely confident." Higher scores denote higher pain self-efficacy. The questionnaire is widely used across various chronic pain conditions and has strong psychometric properties.25 Scores range from 0 to 60. This was prespecified as our primary outcome measure. The Chronic Pain Acceptance Questionnaire40 was used to evaluate chronic pain acceptance. This 20-item survey is composed of 2 factors: 1) "activity engagement": engagement in life activities with pain (11 items), and 2) "pain willingness": willingness to experience pain without trying to engage in unhelpful attempts to control it (9 items). Patients were asked to rate the truth of each item as it applied to them (eg, "My life is going well, even though I have chronic pain."). Items are scored on 7-point scale from 0 "never true" to 6 "always true." Higher scores denote greater levels of pain acceptance. Scores on the "activity engagement" subscale range from 0 to 66; scores on the "pain willingness" subscale range from 0 to 54). The Chronic Pain Acceptance Questionnaire has good psychometric properties28 as well as evidence of clinical utility.40 The Perceived Efficacy in Patient-Physician Interactions21 is a 5-item survey measuring confidence in obtaining medical information and attention to their medical concerns from physicians. Items are scored on a 5-point Likert scale from 1 "not at all confident" to 5 "very confident." The Perceived Efficacy in Patient-Physician Interactions has established validity and reliability in older adults21 and patients with osteoarthritis.35 Pain and pain interference were evaluated using the 3-item Pain Intensity and Interference With Enjoyment of Life and General Activity (PEG).16 Pain intensity was rated on an 11-point numeric rating scale, from 0 "nopain" to 10 "pain as bad as you can imagine." For interference items, patients indicated how much pain interfered with enjoyment of life and with general activity from 0 "does not interfere" to 10 "completely interferes." The PEG total score is the mean of these 3 items, where higher values denote a higher level of pain intensity and interference. The PEG has established reliability and validity in a community and veteran populations with chronic pain and has shown responsiveness to improvement similar to the Brief Pain Inventory.15 The PEG was completed as part of the participant's regular clinical care. Assessments within 2 months of the primary PTSM outcome assessment were used for these analyses. To evaluate satisfaction with pain treatment, participants were asked to choose the number between 0 "extremely dissatisfied" and 10 "extremely satisfied" that best reflected how satisfied they are with the results of their pain treatment, in general.

Study Procedures Consecutive new patients who attended the UW CPR between April 2016 and March 2017 completed a collection of pain-relevant patient-reported outcome questionnaires using PainTracker to facilitate comprehensive multidimensional pain care. All new patients were asked to complete the online questionnaires 1 week before their scheduled appointment. Those who were scheduled for a follow-up appointment at UW CPR and completed the follow-up PainTracker assessment were presented with a question determining interest in the PTSM study. If patients were interested in learning about the study, they were directed to an online information statement outlining the purposes and procedures of the study and given the opportunity to enroll. Patients who chose to not consent at the time were given the options to decide at a later time or obtain more information regarding the study. These patients were then sent a followup e-mail by the research team. Intervention and control subjects were compensated with a $100 gift card for completion of all outcome measures.

A controlled, sequential, nonrandomized study design was used. During the first 6 months of the enrollment period, assessment procedures for the control group were conducted. The control group received treatment as usual in the CPR, with no restrictions on treatment received, including medications, procedures, and sessions with pain psychology, pain psychiatry, and social work that provided support for pain self-management. While control subjects were being assessed, the Web-based PTSM platform for the intervention phase of the study was developed by the multidisciplinary research team, which included investigators from psychiatry, internal medicine, psychology, nursing, social work, computer science, and graphic design. During the second 6 months of the study enrollment period, patients were enrolled in the intervention group. Control as well as intervention subjects were followed for 6 months. There was no restriction on treatments received in either group. The study procedures were reviewed and approved by the institutional review board at UW. Intervention The intervention included exposure, at the patient's discretion, to a Web-based patient empowerment platform on the basis of Acceptance and Commitment Therapy (ACT) principles, as well as phone and text coaching from the research clinicians (P.S.D. and C.T., trained in nursing and social work, respectively). The flow of the study is shown in Fig 1. The PTSM interactive educational modules covered the following topics: module A: "Introduction to PainTracker" is a brief, noninteractive informational module that was presented to the intervention as well as control patients as an introduction to the first PainTracker assessment. Module B: "What is Pain?," explained that pain is important, unpredictable, and complex. It emphasized that all pain is real and important. It also emphasized that pain may get better and worse for unclear reasons. It did not focus on the difference between acute and chronic pain. Education on the complexity of pain used concepts of "injury" versus "alarm," and incorporated some ideas from Explain Pain by Butler and Moseley.5,23 Module C: "Life Navigation System," assisted patients with clarifying values and developing an action plan to improve 1 selected life area (ie, free time, relationships, health and self-care, or work and education). This module was adapted from a treatment manual written by Vowles and Sorrell38 and incorporated the Values Bullseye exercise of Lundgren and colleagues.19 Module D: "Get Rhythm," focused on pacing, mindful breathing, and sleep rhythms. These 3 areas were selected for skill development because they are often core components of behavioral treatments for chronic pain and because of their relevance with the values focus of the intervention. Participants were encouraged to bring some regular rhythm into their lives, particularly as related to engagement in valued living. Module E: "Life Goes On," the final module, focused on scheduling value-based activities and managing pain flares over the longer term. These themes were chosen to emphasize the importance of engagement in value-based activities for sustained recovery.2 Intervention participants were given access to all modules at the outset of the study. They were not forced to complete them on a schedule or in order. The coaches strived to have at least 1 coaching session after the completion of each module.The coaches estimate that patients spent 30 to 40 minutes on each module that they viewed. Module A was especially short and Module B was especially long. Total estimated time for module viewing was 120 to 160 minutes. More precise tracking of viewing time was not possible because of patients' ability to leave the modules open while they attend to other things. Embedded in each of the interactive modules were open-ended and multiple choice questions and tasks, such as "Of all the things that have happened to you since your pain started, what concerns you the most?" or "Create your own action plan." The responses to these module questions were visible to the coaches and were used to guide and tailor the coaching sessions to the individual patient. Coaching sessions occurred in person (14%), over the phone (85%), or by e-mail and text (1%), on an average of 4 occasions (SD = 1.6) depending on participant preference and availability, with a mean duration of 20 minutes (SD = 8.6, range = 2-50 minutes per session). After each individual coaching session, participants were sent an e-mail summary of the recommendations discussed. At study completion, a final note was sent with a summary of key self-management strategies, and encouragement to continue to incorporate them into daily life. The patient coach's general approach within each coaching session was to use open, active listening strategies to establish therapeutic rapport. Coaching sessions were focused on incorporating and engaging participants in the PTSM study educational content. Module content was reviewed and questions or concerns were addressed. Participants were asked to identify 1 to 2 simple and achievable goals on the basis of suggestions in the module, and were guided to identify specific strategies to meet the goal. Efforts were made to redirect conversations from excessive review of pain complaints to values, functioning, goal-setting, and self-care. Questions regarding specific diagnoses or medical therapies were directed to the UW CPR provider. Each week, the team met to discuss 1 or 2 challenging cases, and to provide the research clinicians with supervision. Suggestions for strategies to promote engagement in the study educational content were provided by pain psychiatry and psychology (M.S., K.E.V., R.V.). Brief summaries of the coaching session and customized suggestions for engagement of the patient in pain self-management were provided to the patient's UW CPR provider at their next clinic visit on a printed sheet placed on top of the patient's clinical chart.

Data Analysis Data were analyzed using SPSS version 25 (IBM Corp, Armonk, NY). Descriptive statistics and frequency distributions were calculated for sample characteristics. Independent samples t-tests for continuous variables and χ2 tests for categorical variables were used to evaluate for differences in demographic and clinical characteristics between the control and intervention groups. Adjustments were not made for missing data. A P value of <.05 was considered statistically significant. Generalized estimating equations (GEE) were used to evaluate the effect of the intervention on primary (pain self-efficacy) and secondary (chronic pain acceptance, perceived efficacy in patient-provider interactions, pain intensity and interference, satisfaction with pain treatment) outcomes. GEE is an extension of generalized linear models that allows for the analysis of repeated measures with unknown covariance structure. GEE uses any and all available data that participants provide, even if follow-up data are missing (ie, intent-to-treat analysis). For all models, the main effect of group and time, and the Group × Time interaction were evaluated. For this pilot study,Wald χ2 statistics with P values <.05 for overall model effects were considered statistically significant. For models with significant Group × Time interactions, the main effects of group or time were not reported. For models with only a significant main effect of time, models were rerun without the interaction term to obtain the true main effect. GEE models for the entire study sample and for only those who provided outcome data at all study time points (baseline, 3 months, 6 months) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All new patients receiving care at University of Washington's Center for Pain Relief (UWCPR) and planning ongoing pain care by providers at UWCPR (not one-time consults or procedure patients), with a diagnosis of one or more chronic pain disorders
* *Note: Eligible patients will be invited to participate in the study after completing their second PainTracker pre-UWCPR visit assessment.

Exclusion Criteria:

* Patients attending UWCPR for only a single session or for only evaluation
* Patients participating in 6-week Pain Support Groups at UWCPR or Harborview Medical Center for the duration of the 6-month study
* Unable to read and write English
* Dementia or other significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Sullivan, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Center for Pain Relief, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A controlled, sequential, nonrandomized study design was used. For first 6 months of enrollment, assessment procedures for the control group were conducted, during which the Web-based PTSM platform for the intervention phase of the study was developed. During the second 6 months, patients were enrolled in the intervention group.
Period: Overall Study
Arm/Group | Usual Care | PainTracker Self-Manager
Started | 51 | 48
Completed | 45 | 37
Not Completed | 6 | 11
Not completed — Withdrawal by Subject | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | PainTracker Self-Manager | Total
Number analyzed (Participants) | 51 | 48 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.23 (13.95) | 45.29 (14.34) | 46.29 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 39 | 30 | 69
  Unknown or Not Reported | 9 | 16 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 39 | 30 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 15 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 48 | 99
Pain Self-Efficacy Questionnaire (PSEQ) [Mean (Standard Deviation); unit: score on a scale] — The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item survey that assesses patients' pain self-efficacy, or confidence in their ability to cope with pain and continue activities of daily living. Items are scored on a 7-point scale from 0 "not at all confident" to 6 "completely confident." Total (sum) scores range from 0 to 60, where higher scores denote higher pain self-efficacy.
  score on a scale | 24.74 (12.71) | 24.43 (12.78) | 24.59 (14.10)
Chronic Pain Acceptance Questionnaire (CPAQ) [Mean (Standard Deviation); unit: score on a scale] — The Chronic Pain Acceptance Questionnaire (CPAQ) evaluates chronic pain acceptance. This 20-item survey is composed of 2 factors: 1) "activity engagement": engagement in life activities with pain (11 items), and 2) "pain willingness": willingness to experience pain without engaging in unhelpful attempts to control it (9 items). Participants rate each item on 7-point scale from 0 "never true" to 6 "always true." Subscale (sum) scores range from 0 to 66 for "activity engagement" and 0 to 54 for "pain willingness". Higher scores denote greater levels of pain acceptance.
  score on a scale
    CPAQ - Activity Engagement Subscale | 29.26 (11.55) | 29.48 (11.87) | 29.37 (11.65)
    CPAQ - Pain Willingness Subscale | 20.22 (8.05) | 19.65 (6.91) | 19.94 (7.47)
Perceived Efficacy in Patient-Physician Interactions (PEPPI-5) [Mean (Standard Deviation); unit: score on a scale] — The Perceived Efficacy in Patient-Physician Interactions is a 5-item survey measuring confidence in obtaining medical information and attention to patients' medical concerns from physicians. Items are scored on a 5-point scale from 1 "not at all confident" to 5 "very confident." Total (sum) scores range from 5 to 25, where higher scores denote greater confidence.
  score on a scale | 17.39 (4.76) | 17.83 (4.91) | 17.61 (4.82)
Pain severity, Enjoyment of life interference, General activity interference (PEG) [Mean (Standard Deviation); unit: score on a scale] — Pain and pain interference were evaluated using the 3-item Pain Intensity and Interference With Enjoyment of Life and General Activity (PEG). The pain intensity item was rated on an 11-point numeric rating scale, from 0 "no pain" to 10 "pain as bad as you can imagine." For interference items, patients indicated how much pain interfered with enjoyment of life and with general activity from 0 "does not interfere" to 10 "completely interferes." The PEG total (mean) score ranges from 0 to 10, where higher scores denote greater pain intensity and interference.
  score on a scale | 6.82 (1.95) | 6.99 (1.77) | 6.90 (1.86)
Satisfaction with pain treatment [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to select a number between 0 "extremely dissatisfied" and 10 "extremely satisfied" that best reflected how satisfied they are with the results of their pain treatment, in general. This measure was a single item that ranged from 0 to 10.
  units on a scale | 4.39 (2.62) | 4.15 (2.41) | 4.28 (2.51)

OUTCOME MEASURES:

1. Primary Outcome: Chronic Pain Self-efficacy
Description: Pain self-efficacy questionnaire (PSEQ); scores range from 0 to 60, with higher scores meaning greater self-efficacy (i.e., better outcome)
Time Frame: 3 months and 6 months
Population: Analyzed number from those who provided data at all 3 time points (0, 3 months, 6 months.); published manuscript describes methodology for assessing change over time in outcomes between the two groups (generalized estimating equations), using data from (1) all enrolled participants and (2) only participants who provided data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | PainTracker Self-Manager
Number analyzed (Participants) | 45 | 37
score on a scale
  3 months: number analyzed (Participants) | 42 | 35
  3 months | 27.33 (14.71) | 33.66 (12.28)
  6 months: number analyzed (Participants) | 44 | 35
  6 months | 28.39 (13.68) | 35.57 (12.29)
Statistical Analysis 1: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate improvement in pain self efficacy over time compared to the usual care group; Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis. GEE allows for the analysis of repeated measures with unknown covariance structure and uses all available data that participants provide, even if follow-up data are missing (ie, intent-to-treat analysis). Models for the entire study sample and for only those who provided outcome data at all study time points (0, 3, 6 months; i.e., as treated 'completer' analysis) were evaluated (see Statistical Analysis 2); p < 0.05, Wald χ2 — Wald χ2 p-values < 0.05 considered statistically significant for group x time interactions; Intent-to-treat analysis (full sample)
Statistical Analysis 2: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate improvement in chronic pain self-efficacy over time compared to the usual care group. This analysis was limited to those participants who provided data at each of the study time points ('completer analysis'); Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis; p < 0.05, Wald χ2 — Wald χ2 values < 0.05 considered statistically significant for group x time interactions; Study 'completers' only

2. Secondary Outcome: Chronic Pain Acceptance
Description: Chronic Pain Acceptance Questionnaire with 2 subscales: Activity Engagement and Pain Willingness. Scores on the "activity engagement" subscale range from 0 to 66; scores on the "pain willingness" subscale range from 0 to 54; higher scores denote greater chronic pain acceptance.
Time Frame: 3 months and 6 months
Population: While participants may have provided data at all time points, they may have not provided sufficient data to calculate a score on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | PainTracker Self-Manager
Number analyzed (Participants) | 45 | 37
score on a scale
  CPAQ-Activity Engagement; 3 months: number analyzed (Participants) | 43 | 36
  CPAQ-Activity Engagement; 3 months | 31.05 (11.22) | 36.36 (11.00)
  CPAQ-Activity Engagement; 6 months: number analyzed (Participants) | 44 | 36
  CPAQ-Activity Engagement; 6 months | 32.91 (10.21) | 38.00 (9.62)
  CPAQ-Pain Willingness; 3 months: number analyzed (Participants) | 42 | 36
  CPAQ-Pain Willingness; 3 months | 20.69 (8.98) | 23.06 (7.56)
  CPAQ-Pain Willingness; 6 months: number analyzed (Participants) | 44 | 36
  CPAQ-Pain Willingness; 6 months | 21.00 (8.16) | 23.83 (6.87)
Statistical Analysis 1: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate improvement in chronic pain acceptance - Activity Engagement - over time compared to the usual care group. Note: this questionnaire has 2 subscales, Activity Engagement and Pain Willingness. Intent-to-treat and as treated analyses were conducted for each subscale; Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis. Main effects of group and time, and group × time interactions were evaluated. Models for the entire study sample and for only those who provided outcome data at all study time points (0, 3, 6 months; 'study completers') were evaluated (see Statistical Analysis 2); p = 0.068, Wald χ2 — Wald χ2 p-values < 0.05 considered statistically significant for group x time interaction; Intent-to-treat analysis (full sample)
Statistical Analysis 2: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group by time interaction, such that the PTSM group would demonstrate improvement in chronic pain acceptance - Activity Engagement - over time compared to the usual care group.This analysis was limited to those participants who provided data at each of the study time points ('completer' analysis); Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis; p < 0.05, Wald χ2 — Wald χ2 <0.05 considered statistically significant for group x time interaction; Study 'completers' only
Statistical Analysis 3: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group by time interaction such that the PTSM group would demonstrate improvement in chronic pain acceptance - Pain Willingness - over time compared to the usual care group; Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis; p = 0.173, Wald χ2 — Wald χ2 < 0.05 considered statistically significant for group x time interaction; Intent-to-treat analysis (full sample)
Statistical Analysis 4: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group by time interaction such that the PTSM group would demonstrate improvement in chronic pain acceptance - Pain Willingness - over time compared to the usual care group. This analysis was restricted to those study participants who provided data at each of the study time points ('completer' analysis); Test type: Other — Generalized estimating equations were used to test this hypothesis; p = 0.167, Wald χ2 — Wald χ2 >0.05 considered statistically significant for group x time interaction; Study 'completers' only

3. Secondary Outcome: Patient-physician Interactions
Description: Perceived efficacy in patient-physician interactions (PEPPI). Sum scores range from 5 to 25 with higher scores denoting greater perceived efficacy in patient-physician interactions.
Time Frame: 3 months and 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | PainTracker Self-Manager
Number analyzed (Participants) | 45 | 37
score on a scale
  3 months: number analyzed (Participants) | 43 | 36
  3 months | 17.53 (4.61) | 19.22 (3.89)
  6 months: number analyzed (Participants) | 44 | 36
  6 months | 17.75 (5.23) | 20.03 (5.02)
Statistical Analysis 1: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate improved confidence in patient-provider interactions over time compared to the usual care group; Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis. Main effects of group and time, and group × time interactions were evaluated. Models for the entire study sample and for only those who provided outcome data at all study time points (0, 3, 6 months) were evaluated (see Statistical Analysis 2); p = 0.176, Wald χ2 — Wald χ2 p-values < 0.05 considered statistically significant for group x time interaction; Intent-to-treat analysis (full sample)
Statistical Analysis 2: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate improved confidence in patient-provider interactions over time compared to the usual care group. This analysis was restricted to those study participants who provided data at each of the study time points ('completer' analysis); Test type: Other — Generalized estimating equations were used to test this hypothesis; p = 0.143, Wald χ2 — Wald χ2 < 0.05 considered statistically significant for group x time interaction; Study 'completers' only

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with care process. Note that we elected to evaluate patient satisfaction with their pain treatment in general, as opposed to the PTSM process specifically, in order to compare satisfaction between the study groups. Patient satisfaction was rated on an 11-point rating scale from 0 "extremely dissatisfied" to 10 "extremely satisfied"; higher scores denote higher satisfaction with pain treatment.
Time Frame: 3 months and 6 months
Population: While participants may have provided outcome data at all time points, they may have not provided satisfaction data for this item within 2 months of primary outcome measure collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | PainTracker Self-Manager
Number analyzed (Participants) | 51 | 47
score on a scale
  3 months: number analyzed (Participants) | 45 | 38
  3 months | 5.07 (2.49) | 5.39 (2.47)
  6 months: number analyzed (Participants) | 49 | 39
  6 months | 5.27 (2.88) | 6.36 (2.21)
Statistical Analysis 1: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate improved satisfaction with pain treatment over time compared to the usual care group; Test type: Other — [test comment as in outcome 3, analysis 1]; p < 0.05, Wald χ2 — Wald χ2 p-values < 0.05 considered statistically significant; Intent-to-treat analysis (full sample)
Statistical Analysis 2: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate improved satisfaction with pain treatment over time compared to the usual care group. This analysis was restricted to those study participants who provided data at each of the study time points (i.e., 'completer' analysis); Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis; p < 0.001, Wald χ2 — Wald χ2 < 0.05 were considered statistically significant for the group x time interaction; Study 'completers' only

5. Secondary Outcome: Provider Satisfaction
Description: Provider satisfaction with care process and PTSM
Time Frame: 6 months
Population: While providers were informed of study and coaching progress, we did not formally enroll providers in the study.
Arm/Group | Usual Care | PainTracker Self-Manager
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pain Severity, Enjoyment of Life Interference, General Activity Interference (PEG)
Description: Pain and pain interference were evaluated using the 3-item PEG scale. The pain intensity item was rated on an 11-point numeric rating scale, from 0 "no pain" to 10 "pain as bad as you can imagine." Interference (with enjoyment of life and general activity) were rated from 0 "does not interfere" to 10 "completely interferes." The PEG total (mean) score ranges from 0 to 10, where higher scores denote greater pain intensity and interference.
Time Frame: 3 months and 6 months
Population: While participants may have provided outcome data at all time points, they may have not provided sufficient data for on this scale within 2 months of primary outcome measure collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | PainTracker Self-Manager
Number analyzed (Participants) | 51 | 47
score on a scale
  3 months: number analyzed (Participants) | 34 | 41
  3 months | 6.83 (2.35) | 6.06 (1.93)
  6 months: number analyzed (Participants) | 32 | 38
  6 months | 6.51 (1.94) | 6.06 (1.96)
Statistical Analysis 1: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate greater reductions in pain intensity and interference over time compared to the usual care group; Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis.Models for the entire study sample and for only those who provided outcome data at all study time points (0, 3, 6 months) were evaluated (see Statistical Analysis 2); p = 0.102, Wald χ2 — Wald χ2 p-values < 0.05 considered statistically significant; Intent-to-treat analysis (full sample)
Statistical Analysis 2: Comparison: Usual Care vs PainTracker Self-Manager; We hypothesized that we would observe a group (usual care vs PTSM) by time (0, 3, 6 months) interaction, such that the PTSM group would demonstrate greater reductions in pain intensity and interference over time compared to the usual care group. This analysis was restricted to those study participants who provided data at each time point (as treated, 'completer' analysis); Test type: Other — Generalized estimating equations (GEE) were used to test this hypothesis; p < 0.05, Wald χ2 — Wald χ2 < 0.05 considered statistically significant for group x time interaction; Study 'completers' only

ADVERSE EVENTS:
Time Frame: 6 months (baseline to 6-month follow-up)
Description: The study was low-risk - no forseeable risk for Serious Adverse Events for any of the participants.
Arm/Group | Usual Care | PainTracker Self-Manager
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 0/51 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03045081/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03045081/SAP_001.pdf
  • Informed Consent Form (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03045081/ICF_002.pdf